CLINICAL TRIAL: NCT03866759
Title: European HIV&STI Prevention Network Study
Brief Title: Prospective Observational Cohort HIV & STI Study in Europe
Status: Completed | Type: Observational
Sponsor: Hendrik Streeck (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor-Investigator, Hendrik Streeck, Prof. Dr. med. Hendrik Streeck, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Other Study IDs: STIPnet Study
Record Dates: First submitted 2019-02-15; First posted 2019-03-07 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: HIV Infections; HIV-1-infection; Risk Reduction; Sexual Behavior
Keywords: Sexually Transmitted Infection; HIV Vaccine Trials Network; Pre-exposure prophylaxis
MeSH Terms: conditions — HIV Infections; Risk Reduction Behavior; Sexual Behavior; Sexually Transmitted Diseases | interventions — Prevalence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Blood (Serum, Plasma) Swabs (oral,rectal)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Determine the Incidence and Point Prevalence — Determine the Incidence and Point Prevalence of human immunodeficiency virus (HIV) Infection and the Most Common Sexually Transmitted Infections in Individuals With Sexual Risk Behavior.

SUMMARY:
The University Hospital Essen is sponsoring the Multicenter human immunodeficiency virus (HIV) and sexually transmitted infections Prevention Network Study (STIPnet) which is funded by Janssen, Pharmaceutical Companies of Johnson & Johnson.

STIPnet study is a prospective observational cohort study aiming to determine the incidence and point prevalence of HIV infection and the most common sexually transmitted infections (STIs) in individuals with sexual risk behavior. In addition, the University Hospital Essen will examine whether individuals at risk for HIV and STI infections would retain in such a study (retention rate) and would be willing to participate in potential HIV and STI prevention trials (willingness to participate).

DETAILED DESCRIPTION:
To develop and test novel prevention methods or interventions against sexually transmitted infections (STIs), knowledge is required on whether there are increased rates of transmission in a given population. In order for trials testing new prevention methods to be feasible and affordable, the goal is to define a group at risk where there will be at least an annual 3% incidence of new infections of the respective STI. The group definitions will be based on factors such as gender, age, sexual behavior, economic status and others. However, defining such groups is labor-intensive and costly and often not do-able for vaccine developers and developers of novel prevention/diagnostic methods. Thus, as identification and testing of the most at-risk groups to study these medicinal products is too costly, only a limited number of novel prevention methods are brought into clinical trials. Here the investigators plan to define factors such as behavioral or co-infections associated with individual STIs for potential future prevention trials. Given the increased susceptibility of human immunodeficiency (HIV) infection with STI infections, early diagnosis and treatment of STI is substantial to reduce risk factor of HIV acquisition and to inform individuals about their risk of becoming HIV infected. As STIs are a crucial factor in the scope of an incidence analysis of HIV in men who have sex with men (MSM) and are often underdiagnosed, extensive screening measures are implemented within this study.

Thus, the STIPnet study is building up a platform for effective recruitment, retention and assess important epidemiological patterns and thus, designed as a vaccine preparedness study, to gather information on the most common STIs and prepare sites for potential future vaccine trials. Indeed, several potential HIV&STI vaccines are currently in development.

At-risk volunteers are screened every three months for HIV and other STIs, thereby establishing disease prevalence and incidence in communities that might someday support future vaccine trials. Behavioural data are also collected and participants complete a questionnaire that assesses the willingness to participate in future vaccine studies.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-uninfected as defined as negative HIV-Ab-Elisa, negative HIV viral load or negative HIV Ag-Test at time point of screening.
2. 18-55 years of age
3. Male sex - (at birth, chosen or intersex)
4. Able and willing to give informed consent
5. Able to read and write in local or English language
6. Willing to show identification card
7. Willing to be followed for at least 12 months in the study and undergo study procedures including testing for HIV and receipt of HIV test results
8. Willing to provide contact information for themselves and, if available, one personal contact who would know their whereabouts during the study period
9. Willing to provide information regarding risk behaviors
10. Demonstrates any one of the following risk factors:

    1. reports condomless anal intercourse with at least two unique male partners (unknown HIV status or HIV+ untreated individuals) in the past 24 weeks or
    2. documented history (lab work, physician's note etc) of syphilis, rectal neisseria gonorrhea, mycoplasma genitalium, chlamydia or acute Hepatitis C virus (HCV) infection in the past 24 weeks

Exclusion Criteria:

1. Any significant condition (including medical, psychologic/psychiatric and social) which, in the judgment of the study investigator, might interfere with the conduct of the study or be detrimental to the participant.
2. Prior or concurrent participation in a candidate HIV vaccine study, unless documented placebo recipient.
3. Concurrent participation in investigational HIV treatment or prevention studies (Please note: previous participation is not an exclusion criterion).
4. Employees of the study sites cannot participate but are eligible to participate at a different study site.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men who have sex with Men (MSM) Transgender Men (TGM) Transgender Women (TSW) Intersex
Study Population: The study population will consist of a minimum of 3,300 and a maximum of 3,800 HIV uninfected men who have sex with men (MSM)/Transgender Men (TGW)/Transgender Woman (TGM)/Intersex ages 18-55 years at risk for HIV infection at all study sites. Each participant will be followed for a total of 12 months with assessment of HIV and STI status and risk behavior conducted at screening/enrollment, three months (V1), six months (V2), nine months (V3), and twelve months (V4). It is anticipated that total accrual will take until LPI is enclosed. It is estimated that a total of max. 4,540 participants will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 3593 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Choice of a cohort of volunteers at-risk for HIV and other STIs | Through study completion, an average of 2 years
  Participants will receive questionnaires. The group definitions will be based on factors such as gender, age, education, sexual behavior, economic status, pre- and post-exposure prophylaxis and others. Descriptive statistics will be generate to choose a cohort of volunteers at-risk for HIV and other STIs.
Relationship between STIs and certain behavior and risk of HIV infection | Through study completion, an average of 2 years
  Participants will receive a questionnaire about behavior and risk of HIV infection. Descriptive statistics will be generate to summarize the relationship between STIs and HIV infection.
Incidence of HIV and other STIs in a cohort of individuals at risk for HIV and other STI infections | Through study completion, an average of 2 years
  Descriptive statistics will be generated to summarize incidence (as measured as new HIV and STI infections occurring during the study period) HIV and STI infections. The power calculation targets a 3% incidence rate per year.

SECONDARY OUTCOMES:
Prevalence of HIV and other STIs in a cohort of individuals at risk for HIV and other STI infections | At screening (until last participant is included), an average of 1 year
  Descriptive statistics will be generated to summarize prevalence (as measured as HIV and STIs positive cases during screening visit) HIV and STI infections. Baseline HIV and STI prevalence will be defined as the number of HIV or STI infected individuals identified at screening divided by the total number of individuals who are screened for HIV or STI.
  Once enrollment is completed, baseline HIV or STI prevalence will be calculated.
Co-occurence of STIs and HIV | Through study completion, an average of 2 years
  Analysis of laboratory and other testing results. Descriptive statistics will be generated to evaluate co-occurence of STIs and HIV.
Retention rates for prospective prevention studies for individuals at risk for HIV and STI infections. | Through study completion, an average of 2 years
  The primary assessment of retention will be conducted assuming a binomial distribution and individuals will be considered retained at 12 months if they complete the final study visit. Retention will also be estimated with 95% CI for each study visit. A summary of participant attendance and loss to follow-up will be made every 3 months to monitor the retention rate by site, and to help ensure that the overall 12-month retention rate of the study visit will be no less than 85%.
Willingness to participate in future clinical trials, such as those of candidate vaccines through questionnaire | At enrollment (day 0, can be same day as screening day) and at visit 4 (visit 4 is day 364)
  Willingness to participate in vaccine trials will be estimated assuming a binomial distribution. Factors associated with willingness to participate in vaccine trial will be evaluated using logistic regression models
Attitudes regarding HIV and STI prevention methods | At screening, at visit 1, 2, 3, 4 (visit 1 is day 84, visit 2 is day 168, visit 3 is day 252 and visit 4 is day 364)
  Attitudes regarding PrEP will be evaluated using descriptive statistics and questionnaires. Behavioral questionnaire over time will be assessed by frequency tables and bar graphs.
Incidence between individuals at risk for HIV and STI infections across sites and countries | Through study completion, an average of 2 years
  Descriptive statistics will be generated to summarize incidence (as measured as new HIV and sexual transmitted infections occurring during the study period) HIV and STI infections. Data may be compared across sites for comparison and evaluation of factors impacting incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Streeck, Prof. Dr., Principal Investigator — Institute for HIV Research
Locations (15):
- France (5):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Hôpital de la Croix-Rousse, Lyon
  - Hospital Saint Louis, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Antoine, Paris
- Semmelweis University, Budapest, Hungary
- Italy (3):
  - Hospital Maggiore Policlinico, Milan
  - Hospital San Raffaele, Milan
  - National Institute for Infectious Diseases L. Spallanzani, Rome
- Poland (4):
  - Centrum PrEP Gdańsk, Gdansk
  - Pomeranian Medical University, Szczecin
  - Chmielna Express Warsaw, Warsaw
  - Center for Prevention and Treatment of Infectious Diseases and Addiction Treatment, Wroclaw
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Vall d'Hebron Research Institute, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
The study collaborators recognize the importance of disseminating scientific and medical study data as soon as the study data sets are complete and analysed; therefore, the study leadership would encourage their presentation, discussion and publication at seminars or conferences (national, regional and international) and in reputable scientific journals in open access. All publications resulting from this study will be cleared through the collaborating partners to the study. Anonymous data can be obtained upon request to the PI of the study.Confidentiality of participants will be maintained by the fact that no individual results will be reported or published, only group/aggregate results. Data collected during the trials that underlie the results presented in scientific publications will be shared. Distribution of study data must be always approved by the scientific steering committee of the study and final approval needs to be obtained by the PI.
Time Frame: After publication. No end date
Access Criteria: Researchers who would like to access the data after completion of trial should provide a written request to studien@hiv-forschung.de